CLINICAL TRIAL: NCT03007589
Title: Natural Sunlight Protection and Simulated Sunlight Protection Offered by Sunscreens and Fabrics
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Protection Foundation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPF-2014-001
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Sunburn; Sun Damaged Skin; Overexposure to Sun Rays
Keywords: erythema; persistent pigment darkening; sunburn; suntan
MeSH Terms: conditions — Sunburn; Erythema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Location (Other): Location and Intensity of Exposure to Sunlight otc sunscreens sun protection fabrics optical filters
  Interventions: Drug: otc sunscreens; Other: sun protection fabrics; Other: Optical Filters
- Single Duration or SPF Test (Other): Single exposure of interventions or multiple exposures of interventions (SPF or PPD-PF tests) otc sunscreens sun protection fabrics optical filters
  Interventions: Drug: otc sunscreens; Other: sun protection fabrics; Other: Optical Filters

INTERVENTIONS:
Drug: otc sunscreens — Sunscreens of various SPF levels and ingredients
  Other Names: 30 SPF Broad Spectrum Sunscreen; 40 SPF Broad Spectrum Sunscreen; 45 SPF Broad Spectrum Sunscreen; 50 SPF Broad Spectrum Sunscreen; 60 SPF Broad Spectrum Sunscreen; 100 SPF Broad Spectrum Sunscreen; 110 SPF Broad Spectrum Sunscreen; Sunscreen Standard P2 15 SPF; Sunscreen Standard S2 12 UVA-PF; Sunscreen Standard P1 4 SPF; 70 SPF Broad Spectrum Sunscreen; 85 SPF Broad Spectrum Sunscreen; Reference Standard Sunscreens at various SPF levels
Other: sun protection fabrics — fabrics
  Other Names: 100+ SPF Broad Spectrum Fabric Solumbra; 30+ SPF Broad Spectrum Fabric Solumbra
Other: Optical Filters — Optical band pass or long pass filters or surfaces/mirrors used in solar simulators
  Other Names: Pass Through Glass

SUMMARY:
The purpose of this study is to assess how human skin reacts and how sunscreens and sun protection fabrics protect in natural sunlight compared to their labeled claims, indoor testing methods (existing or modified) and instructions.

DETAILED DESCRIPTION:
To evaluate the difference in the level of erythema and persistent pigment darkening sun protection following a single period of natural sunlight exposure or laboratory solar simulator exposure afforded by application of sunscreens, use of fabrics, and use of pass through glass filters.

ELIGIBILITY:
Inclusion Criteria:

1. Fitzpatrick Type I, II, III, IV or V type skin.
2. Must be able to be exposed to natural sunlight for up to 4 hours in a prone position
3. Able to read, write, speak and understand the English language.
4. Has personally read, signed, and dated the Informed Consent Form (including HIPAA disclosure) and Photograph Release
5. Generally in good health based on medical history reported by the subject
6. Healthy male or female subjects with no history or evidence of clinically relevant medical disorder, as determined from a brief medical history interview.
7. Willing and able to follow the study instructions, including:

   * Remain outdoors exposed to the sun or in the laboratory for up to 4 hours on Day 1 during the study with exposed skin on back protected by sunscreens and fabrics
   * Apply the specific sunscreens and fabrics to designated sites on the back and lie motionless.
   * No visual signs of recent sun exposure to the back.
   * No sunscreens or lotions recently used on the back.
   * Attend scheduled visits and intend to successfully complete the study
   * Stay out of the sun or stay indoors from sun exposure until after observation on Day 2.
   * Women are discouraged from using a bra that applies pressure to the skin site areas that may make it difficult to assess erythema or PPD on Day 2.
   * Refrain from using other sunscreen products or tanning bed use during the duration of the study.

Exclusion Criteria:

1. Individuals with known allergies or sensitivities to sunscreens or any ingredient contained in the test products or common topical skincare products, including adhesives.
2. Perceptible erythema, PPD on the back as determined by the PI or designee.
3. Women known to be pregnant or nursing.
4. Individuals with any disease or condition of the skin (e.g., active [i.e. flaring] eczema or psoriasis, skin cancer, atypical nevus, polymorphic light eruption (PMLE), porphyria, systemic lupus erythematous (SLE), xeroderma pigmentosa (XP)) that could interfere with the study or increase risk to the subject.
5. Individuals with self-reported UNCONTROLLED metabolic conditions, such as diabetes, hypertension, hyper/hypothyroidism, hypercholesterolemia
6. Subjects who are taking medication for chronic conditions that may make a subject more sun sensitive (e.g., Tetracyclines, antifungals, certain diuretics, etc.)
7. Skin diseases on tested sites (e.g., photosensitivity disorders, etc.), which may influence the outcome of the study
8. An individual who has any condition which in the PI's judgment makes the candidate an inappropriate subject for study participation
9. Individuals with a condition or situation which, in the PI's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
10. Individual viewed by the PI as not being able to complete the study

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Erythema | 16-24 hours post exposure to natural sunlight
  • Erythema was assessed using a scale of 0 = no perceptible sun induced skin reaction, 1 = perceptible erythema but spotty or without clear borders (<1 MED); 2 = minimal erythema over the entire site with distinct borders (1 MED reaction); 3 = more than minimal; 4 = a serious erythema; and 5 = edema and blisters.
  Determination made by blinded evaluator on-site or using chroma-meter and photographs.
Persistent Pigment Darkening (PPD) | 16-24 hours post exposure to natural sunlight
  Persistent Pigment Darkening was assessed using a scale of 0 = no perceptible sun induced skin reaction, 1 = perceptible but spotty or without clear borders (<1 MPPDD); 2 = minimal PPD over the entire site with distinct borders (1 MPPDD reaction); 3 = more than minimal; 4 = a serious erythema; and 5 = edema and blisters
  Determination made by blinded evaluator on-site or using chroma-meter and photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Hughes, MBA, Principal Investigator — Sun Protection Foundation
Locations (5):
- United States (3):
  - Sun Protection Foundation, San Diego, California
  - Sun Protection Foundation, Waimea, Hawaii
  - Sun Protection Foundation, Seattle, Washington
- Sun Protection Foundation, Santiago, Chile
- Sun Protection Foundation, Arequipa, Peru

IPD SHARING:
Plan to Share IPD: No